CLINICAL TRIAL: NCT06388759
Title: A Phase Ib Study of TQ05105 Tablets for the Treatment of Intermediate and High Risk Myelofibrosis Refractory/Relapsed/Intolerant to Ruxolitinib
Brief Title: TQ05105 Tablet for Myelofibrosis Treatment in Ruxolitinib-Resistant or Intolerant Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-Ib-03
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 Tablets (Experimental): TQ05105 Tablets，28 days as a treatment cycle.
  Interventions: Drug: TQ05105 Tablets

INTERVENTIONS:
Drug: TQ05105 Tablets — TQ05105 Tablets is a Janus kinase 1 (JAK1) and Janus kinase 2 （JAK2） Inhibitor

SUMMARY:
This is an open, single-arm, multi-center clinical study designed to evaluate the efficacy of TQ05105 Tablets in patients with intermediate-risk and high-risk myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participated in this study, signed informed consent forms, and demonstrated good compliance；
* Age: 18 or older (when signing the informed consent form); Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 2; Life expectancy ≥ 24 weeks;
* Patients diagnosed with Primary myelofibrosis (PMF), post polycythemia vera myelofibrosis (post-PV MF), or post essential thrombocythemia myelofibrosis (post-ET MF);
* According to the dynamic international prognostic scoring system (DIPSS), patients with intermediate or high risk of bone marrow fibrosis were evaluated;
* Patients with poor efficacy or intolerant of Ruxolitinib;
* Spleen enlargement;
* Peripheral blood primary cells and bone marrow primary cells were ≤10%;
* No growth factor, colony stimulating factor, thrombopoietin or platelet transfusion was received within 2 weeks before the examination, and the blood routine indexes met the requirements within 7 days before the first administration;
* The Main organ function is normal;
* Men and women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study. Serum human chorionic gonadotrophin（HCG）test is not negative within 7 days before the first administration and must be non-lactating patients.

Exclusion Criteria:

* Patients who have previously received allogeneic stem cell transplantation, or received autologous stem cell transplantation within 3 months before the first administration, or recently planned stem cell transplantation;
* Previous treatment with JAK inhibitors(except ruxolitinib);
* Patients who have previously undergone splenectomy, or received splenic radiotherapy within 6 months before the first administration;
* Other malignancies within 3 years prior to first administration or currently present;
* Patients with multiple factors (such as inability to swallow, postoperative gastrointestinal resection, acute and chronic diarrhea, intestinal obstruction, etc.) affecting oral or absorption of drugs;
* The non-hematological toxicity caused by previous treatment did not return to grade≤1;
* Major surgical treatment or significant traumatic injury within 4 weeks prior to first administration;
* Presence of congenital bleeding disorder and congenital coagulopathy;
* Patients who had arterial/venous thrombosis events within 6 months before the first administration;
* Have a history of mental drug abuse, or have a mental disorder;
* Active or uncontrolled severe infection;
* Active hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection and HCV RNA positive;
* Patients with ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia, QT interval prolongation and ≥ grade 2 congestive heart failure;
* Unsatisfactory blood pressure control despite standard therapy;
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Patients newly diagnosed with pulmonary interstitial fibrosis or drug-related interstitial lung disease within 3 months before the first administration;
* Patients with a history of immunodeficiency disease or organ transplantation;
* Patients with epilepsy requiring treatment;
* Use of any MF medications, any immunomodulators, androgens, any immunosuppressive agents, erythropoietin, aspirin > 100 mg/day within 2 weeks prior to first administration;
* Patients who have received Chinese patent medicines with anti-tumor indications specified in the approved drug package insert of China National Medical Products Administration (NMPA) within 2 weeks before the first administration;
* Patients with uncontrolled pleural effusion, pericardial effusion or ascites;
* There was a history of attenuated live vaccine inoculation within 4 weeks before the first administration, or attenuated live vaccine inoculation was planned during the study period;
* People with known hypersensitivity to the study drug and excipients;
* Patients diagnosed as active autoimmune diseases within 2 years before the first administration;
* Those who participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first administration;
* According to the judgment of the investigators, some situations seriously endanger the safety of the subjects or affect the subjects to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Spleen volume reduction (SVR35)≥35% from baseline | up to 24 weeks
  The proportion of subjects with spleen volume reduction ≥35%from baseline at the end of treatment at week 24.

SECONDARY OUTCOMES:
Optimum effective rate | up to 120 weeks
  The proportion of subjects with at least one spleen volume measurement of ≥ 35% reduction against the baseline.
Onset time of splenic response | up to 120 weeks
  The time interval from the first administration to the date when the spleen volume was reduced by ≥ 35 % from the baseline.
Duration of maintenance of spleen response (DoMSR) ≥35% reduction | up to 120 weeks
  The time between the date when the spleen volume reduction ≥ 35% from baseline for the first time and the date when the spleen volume reduction < 35% from baseline.
Myeloproliferative neoplasm- Symptom Assessment Form- Total Symptom Score (MPN-SAF TSS) : ≥ 50% Reduction from Baseline | up to 24 weeks
  The proportion of subjects whose total symptom score on the Myeloproliferative Neoplasia Symptom Assessment Form-Total Symptom Score (MPN-SAF TSS) scale decreased by at least 50% compared to baseline. MPN-SAF-TSS is an effective tool for evaluating the disease burden in patients with myeloproliferative neoplasms. A higher score indicates more severe symptoms in patients. Each symptom is scored according to its severity, ranging from no symptoms (0 points) to the most severe (10 points), with a total of 10 levels. The sum of the scores for these 10 symptoms constitutes the MPN-SAF-TSS score.
The total symptom score of MPN-SAF TSS decreased compared with baseline | up to 120 weeks
  The total symptom score of MPN-SAF TSS decreased compared with baseline.
Progression-free survival (PFS) | up to 120 weeks
  The time interval from the first medication to the date of the occurrence of any of the following events, whichever occurs first: (1) Spleen volume increased by≥25% compared with the screening period ; (2) Death caused by any cause.
Leukemia free survival (LFS) | up to 120 weeks
  The time interval from the first medication to the occurrence of any of the following events, whichever comes first: ① The date on which the first bone marrow smear displays ≥20% blast cells; ② The first instance where the peripheral blood smear displays ≥20% blasts with an absolute blast count of ≥1×10^9/L, which persists for at least two weeks; ③ Death caused by any reason.
Overall Survival (OS) | up to 120 weeks
  OS is defined as the time from the first time the subject received treatment to death due to any cause.
Incidence of adverse events (AEs) | baseline up to 120 weeks
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Severity of AEs | baseline up to 120 weeks
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug, evaluated according to the CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Union Hospital Tongji College Huazhong University of Science And Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Hong M, Ding D, Zhang M, Gao S, Song L, Wu D, Lao S, Yu D, Chang C. A first-in-class JAK/ROCK inhibitor, Rovadicitinib in patients with myelofibrosis who were refractory or relapsed or intolerant to Ruxolitinib: A single-arm, multicenter, open-label, phase Ib study. Eur J Pharmacol. 2025 Oct 15;1005:178032. doi: 10.1016/j.ejphar.2025.178032. Epub 2025 Aug 5. PMID 40752760